CLINICAL TRIAL: NCT05401435
Title: Reliability of Measuring Blood Pressure With a Smartwatch
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Czech Technical University in Prague (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NIBPsmartwatch22
Record Dates: First submitted 2022-05-23; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-06

CONDITIONS: Blood Pressure; Heart Rate
Keywords: blood pressure measurement; heart rate measurement; smartwatch
MeSH Terms: interventions — Heart Rate

STUDY DESIGN:
Intervention Model Description: Two measuring devices are active simultaneously during single measurement of blood pressure and heart rate on each participant. Measurements are repeated 2 times a day for 28 days. The functioning of two measuring devices is compared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood pressure and heart rate measurement (Experimental): Resting blood pressure and heart rate measurement regularly one value in the morning and evening for 28 days. The volunteer measures the parameters simultaneously on both devices (smartwatch and digital tonometer). In total, each participant will undergo this measurement 56 times.
  Interventions: Other: Resting measurement of blood pressure and heart rate

INTERVENTIONS:
Other: Resting measurement of blood pressure and heart rate — Simultaneous blood pressure and heart rate measurement every morning and evening during the duration of the experiment (28 days).

SUMMARY:
The aim of this study is to verify the long-term accuracy of blood pressure and heart rate measurements by Samsung smartwatches between two consecutive calibrations compared to a standard digital tonometer used in clinical practice and for home measurement of these vital parameters.

DETAILED DESCRIPTION:
Recently, smartwatches can measure a wide range of biological signals, including heart rate and blood pressure. The short-term reliability of blood pressure measurements after the required calibration has been studied, but long-term reliability is still a question. The aim of the project is to experimentally evaluate the reliability of long-term blood pressure measurement with a Samsung smart watch between two consecutive calibrations over a period of 28 days in comparison with a digital tonometer (Omron) approved as a medical device. Volunteers will measure blood pressure and heart rate manually twice a day from a smartwatch and a digital tonometer simultaneously. The agreement of the measurements of both devices will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* any acute illness
* pregnancy
* severe cardiovascular conditions
* severe asthma or other severe respiratory conditions
* diabetes
* hypotension or hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-05-04 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in long-term similarity of blood pressure measurements from two devices between two consecutive calibrations | 28 days
  The long-term agreement of systolic and diastolic blood pressure measurements of both monitoring devices between two consecutive smartwatch calibrations will be evaluated. This means that we evaluate the changes in the similarity of measured blood pressures over a period of 28 days.
Change in long-term similarity of heart rate measurements from two devices | 28 days
  The long-term agreement of heart rate measurements of both monitoring devices will be evaluated. This means that we evaluate the changes in the similarity of measured heart rates over a period of 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Barbora Nezpevakova, Bc., Principal Investigator — Czech Technical University in Prague; Veronika Rafl Huttova, MSc, Principal Investigator — Czech Technical University in Prague; Martin Rozanek, PhD, Principal Investigator — Czech Technical University in Prague; Jakub Rafl, PhD, Principal Investigator — Czech Technical University in Prague
Locations (1):
- Faculty of Biomedical Engineering, Czech Technical University in Prague, Kladno, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Helmond N, Freeman CG, Hahnen C, Haldar N, Hamati JN, Bard DM, Murali V, Merli GJ, Joseph JI. The accuracy of blood pressure measurement by a smartwatch and a portable health device. Hosp Pract (1995). 2019 Oct;47(4):211-215. doi: 10.1080/21548331.2019.1656991. Epub 2019 Aug 26. PMID 31423912